CLINICAL TRIAL: NCT03554590
Title: Effectiveness of Carbohydrate Counting on Glycaemic Control in T1DM Patients
Brief Title: DM1, Effects of Carbo-Counting on Glycemic Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Emanuela Orsi, Head of DIabetology, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM1cc
Record Dates: First submitted 2017-03-03; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: carbohydrate counting; insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carbo-counters (Experimental): carbohydrate counting: patients attending a structured carbohydrate-counting training and practicing this tecnique to manage insulin therapy
  Interventions: Behavioral: carbohydrate counting
- control group (Active Comparator): insulin therapy according to standard care. patients who don't practice carbohydrate-counting to manage insulin therapy
  Interventions: Behavioral: insulin therapy according to standard care

INTERVENTIONS:
Behavioral: carbohydrate counting — patients will attend a 5 meetings-structured training to learn how to manage their insulin therapy depending on the amount of carbohydrates contained in foods
  Arms: carbo-counters
Behavioral: insulin therapy according to standard care — patients will not manage their insulin therapy depending on the amount of carbohydrates contained in foods, but will follow a fix basal bolus scheme
  Arms: control group

SUMMARY:
Carbohydrate counting is the most effective meal-planning strategy in type 1 diabetes (T1DM) to optimize insulin therapy. However, it may lead to weight gain and unhealthy eating habits. This study aims to compare glycemic control parameters, anthropometric measurements and dietary lifestyle in T1DM patients who practice CHO-counting, after attending a structured course to learn how to manage this tecnique, vs a control Group, in a follow up period of 2 years.

DETAILED DESCRIPTION:
patients with type 1 DM will be enrolled in the study. patients in the intervention group will attend a 5-lessons training to learn how to manage insulin therapy depending on the amount of carbohydrates in their meals, patients in the control group will be follow according to the the standard care. after the follow up period glycometabolic, anthropometric parameters and dietary lifestyle changes will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes mellitus
* insulin therapy
* HbA1c from 5.5 to 10%

Exclusion Criteria:

* pregnancy
* celiac disease
* hepatic impairment
* chronic renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
glycemic control | 2 years
  HbA1c

SECONDARY OUTCOMES:
anthropometric parameters: BMI | 2 years
  variations in body mass index (BMI: units kg/m2), weight and height will be combined to report BMI in kg/m^2
anthropometric parameters: WAIST AND HIP CIRCUMFERENCE | 2 years
  variations in waist and hip circumference (units: cm)
anthropometric parameters: BIOIMPEDENTIOMETRIC PARAMETERS | 2 years
  fat mass and free fat mass (units: % of total mass)
dietary lifestyle | 2 years
  variations in intake of simple sugars, animal protein rich foods, saturated fats and cholesterol, UDM: grams/die. All the informations will be collected using 5days food diaries, completed by the patients.
glucose variability: mean and standard deviation of self monitoring blood glucose (SMBG) | 2 YEARS
  mean and standard deviation of self monitoring blood glucose (SMBG), data collected from glucometers, units: mg/dl
glucose variability: incidence of hypoglycaemia | 2 YEARS
  incidence of hypoglycaemia (SMBG < 70 mg/dl), units: n° episodes/week

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Orsi, Principal Investigator — FOndazione IRCCS Ca' Granda Opedale Maggiore Policlinico Milano
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No